CLINICAL TRIAL: NCT00912080
Title: Utilisation of Genomic Signature as Decision-making for Adjuvant Treatment of Breast Cancer: A Prospective Cohort Study.
Brief Title: Utilization of Genomic Signature as Decision-making for Adjuvant Treatment of Breast Cancer
Acronym: SA02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SA02/IPC 2006-003
Record Dates: First submitted 2009-05-29; First posted 2009-06-03 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: genomic signature; lymph nodes; no metastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- good signature (Experimental): Patients who have a "good signature" for the genomic analysis. They will receive the standard chemotherapy.
  Interventions: Genetic: genomic signature

INTERVENTIONS:
Genetic: genomic signature — genomic signature analysis

SUMMARY:
Method: This multicentric prospective cohort is composed of patients with no metastatic breast cancer selected by tumor's genomic analysis and treated by chemotherapy with Anthracycline without Taxanes (6 cycles of FEC 100).

The patient can be included before or after the surgery and a written consent must be signed for the proteomic and genomic analysis of the tumor.

Patients who have a "good signature" for the genomic analysis will receive the standard chemotherapy.

Primary objective:

* To compare metastasis free survival at 5 years in a cohort of patients with no metastatic breast cancer, who are selected by their genomic profile of the tumor and received a standard chemotherapy containing Anthracycline, with result of retrospectives studies.

Secondary Objectives:

* Overall survival.
* Creation of a circuit (transport-extraction-genomic analysis-result) which allows the beginning of the chemotherapy within 6 weeks following the primary surgery.
* Histological and seric proteomic exploratory studies.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 70
* Patient with life condition < 2 (WHO scale)
* One-sided breast adenocarcinoma with a histological evidence (all type)
* Clinical presentation which allowed a complete surgery with healthy limits
* Absence of metastasis detectable at clinical examination or radiology
* Histological evidence for homolateral axillary ganglionic invasion, whatever is the number of node invaded (N > 1)
* The beginning of the chemotherapy within 6 weeks following the primary surgery

Exclusion Criteria:

* All metastatic affect
* Tumor classed >= T4a: cutaneous invasion, deep adherence, inflammatory breast
* All chemotherapy, hormonotherapy or radiotherapy before surgery
* Tumoral residue not removed
* Any suspect clinic or radiologic lesion, in the contralateral breast, which is not controlled
* History of invasive neoplasm, mammary or other (except in situ carcinoma of cervix uteri and epithelioma)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2007-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Estimation of metastasis free survival at 5 years of the patients who had a good genomic signature. The metastasis free survival is defined by the time between the histological diagnosis of the breast cancer and the apparition of the first metastasis. | 5 years

SECONDARY OUTCOMES:
Time between collection for the genomic signature study and the beginning of the chemotherapy. | 6 weeks
Seric and histological proteomic exploratory studies with SELDI-TOF MS to: search correlation with histo-clinical or/and molecular parameter and to identify one or few proteic signature with a prognosis value. | 6 weeks
Overall survival. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc EXTRA, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (4):
- France (4):
  - Centre Léon BERARD, Lyon
  - Institut PAOLI-CALMETTES, Marseille
  - Centre Antoine LACASSAGNE, Nice
  - Chu Font-Pre, Toulon

REFERENCES:
- See also: official site of the sponsor — http://www.institutpaolicalmettes.fr/